CLINICAL TRIAL: NCT02196623
Title: Hypoxia and Aerobic Exercise Interactions in Age-related Metabolic Muscle Dysfunction
Brief Title: Hypoxia and Exercise in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA 7037/2-1
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2017-08

CONDITIONS: Elderly Persons

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxic Exercise (Experimental): Supervised, progressive aerobic exercise for 8 weeks under hypoxic conditions
  Interventions: Other: Hypoxic exercise
- Normoxic exercise (Sham Comparator): Supervised, progressive aerobic exercise for 8 weeks under normoxic conditions
  Interventions: Other: Normoxic Exercise

INTERVENTIONS:
Other: Hypoxic exercise — Supervised, progressive aerobic exercise program for 8 weeks under hypoxic conditions
  Arms: Hypoxic Exercise
Other: Normoxic Exercise — Supervised, progressive aerobic exercise program for 8 weeks under normoxic conditions
  Arms: Normoxic exercise

SUMMARY:
Ageing is the primary risk factor for most chronic diseases including type 2 diabetes mellitus. Sarcopenia and muscular mitochondrial dysfunction with aging are crucial mechanisms leading to decreased exercise tolerance and worsened insulin sensitivity. Thus, metabolic disease and frailty, which limits physical mobility as well as quality of life, share common cellular mechanisms.

The investigators will test the hypothesis that a combination of normobaric hypoxia and exercise training elicits a synergistic effect on age-associated metabolic skeletal muscle dysfunction and the investigators will address the molecular mechanisms. In a randomized clinical study, the investigators will compare normoxic and hypoxic training conditions in elderly subjects. Outcome measures will focus on whole body insulin sensitivity and mitochondrial responses in skeletal muscle before and after the 8-week training intervention.

ELIGIBILITY:
Inclusion Criteria:

* 55 to 75 years of age
* body mass index: 20 - 35 kg/m2
* weight stable during last 6 months before screening (weight change < 2% body weight)
* HOMA-index of insulin resistance ≥ 2 to 4 units

Exclusion Criteria:

* more than 1 hour of scheduled exercise training per week
* known diagnosis of type 2 diabetes or measured HbA1c > 6,5%
* known drug or alcohol abuse
* any contraindication to perform exercise training
* acute or chronic infections
* increased bleeding risk by history, INR > 1,3, use of anticoagulants

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | At baseline and after 8 weeks
  Insulin sensitivity is assessed via the hyperinsulinemic euglycemic glucose clamp and expressed as the glucose infusion rate (GIR) in ml

SECONDARY OUTCOMES:
Maximum oxygen uptake | At baseline and after 8 weeks
  Maximum oxygen uptake is measured during an incremental exhaustive exercise test and is expressed in ml/min/kg
Mitochondrial number | At baseline and after 8 weeks
  Mitochondrial number and selected gene expression assessed from muscle biopsies from the vastus lateralis.
Fat and carbohydrate oxidation during exercise | At baseline and after 8 weeks
  Fat and carbohydrate oxidation during exercise is assessed during an incremental exercise test by measurements of gas exchange and expressed as g/min
Body fat and body fat free mass | At baseline and after 8 weeks
  Measured via by air-displacement plethysmography (ADP) and expressed in kg
Health related quality of life | At baseline and after 8 weeks
  Assessed using the short form 36 (SF-36) questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sven Haufe, Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] Hein M, Chobanyan-Jurgens K, Tegtbur U, Engeli S, Jordan J, Haufe S. Effect of normobaric hypoxic exercise on blood pressure in old individuals. Eur J Appl Physiol. 2021 Mar;121(3):817-825. doi: 10.1007/s00421-020-04572-6. Epub 2020 Dec 23. PMID 33355713
- [Background] Chobanyan-Jurgens K, Scheibe RJ, Potthast AB, Hein M, Smith A, Freund R, Tegtbur U, Das AM, Engeli S, Jordan J, Haufe S. Influences of Hypoxia Exercise on Whole-Body Insulin Sensitivity and Oxidative Metabolism in Older Individuals. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5238-5248. doi: 10.1210/jc.2019-00411. PMID 30942862